Version: 1.2

## The Ohio State University Combined Consent to Participate in Research and HIPAA Research Authorization

**Study Title:** Pilot study of Tislelizumab (BGB-A317) in recurrent mismatch repair deficient endometrial cancer and the effect on the tumor microenvironment

Principal Investigator: Floor J Backes, MD

Sponsor: BeiGene, Ltd.

- This is a consent form for research participation. It contains important
  information about this study and what to expect if you decide to participate.
  Please consider the information carefully. Feel free to discuss the study with
  your friends and family and to ask questions before making your decision
  whether or not to participate.
- Your participation is voluntary. You may refuse to participate in this study. If you decide to take part in the study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your usual benefits. Your decision will not affect your future relationship with The Ohio State University. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status.
- You may or may not benefit as a result of participating in this study.
   Also, as explained below, your participation may result in unintended or harmful effects for you that may be minor or may be serious depending on the nature of the research.
- You will be provided with any new information that develops during the study that may affect your decision whether or not to continue to participate. If you decide to participate, you will be asked to sign this form and will receive a copy of the form. You are being asked to consider participating in this study for the reasons explained below.

#### **Key Information About This Study**

The following is a short summary to help you decide whether or not to be a part of this study. More detailed information is listed later in this form.

There is an urgent need for new and improved treatment strategies for recurrent endometrial cancer, and methods to identify which patients will benefit from these therapies.

Your tumor has been tested, and is mismatch repair deficient (dMMR). DNA mismatch repair (MMR) is a system for recognizing and repairing DNA errors and damage. You may have acquired this over the course of your life, but in 2-3% of


endometrial cancers this may be due to a hereditary disease called Lynch Syndrome (previously called hereditary nonpolyposis colorectal cancer or HNPCC). Tumors that have evidence of mismatch repair deficiency tend to be more sensitive to immunotherapy. However, immunotherapy is currently only approved for endometrial cancer if the cancer has come back after receiving chemotherapy.

Tislelizumab is an experimental drug. This means that it has not been approved for use by the regulatory agencies (FDA) in the US, but it has been approved in China. Tislelizumab is a monoclonal antibody acting on a protein called Programmed Cell Death 1 (PD-1). In this study, we would like to study how a new immunotherapy (tislelizumab (BGB-A317) works for patients who have not yet received chemotherapy and how the tumor and the immune system respond to treatment. To study this, you will have 2-3 biopsies of your tumor during the study and you will have extra blood samples collected. You will received immunotherapy through a vein every 3 weeks and you will have imaging with CT scans every 3 cycles (every 9 weeks) to see how well the treatment is working. If it does not go away after 3 treatments we will add carboplatin and paclitaxel if you have not had this before, to try to make treatment work better. You can stop treatment at any time. The most likely side effects from immunotherapy are mild and include diarrhea, fever, fatigue, cough, but it can also affect other organs like bowel, kidney, heart, thyroid, lungs, eyes, and other organs. You will be closely monitored for side effects of treatment.

## 1. Why is this study being done?

There is an urgent need for new and improved treatment strategies for recurrent endometrial cancer, and methods to identify which patients will benefit from these therapies.

Your tumor has been tested, and is mismatch repair deficient (dMMR). DNA mismatch repair (MMR) is a system for recognizing and repairing DNA errors and damage. You may have acquired this over the course of your life, but in 2-3% of endometrial cancers this may be due to a hereditary disease called Lynch Syndrome (previously called hereditary nonpolyposis colorectal cancer or HNPCC). Tumors that have evidence of mismatch repair deficiency tend to be more sensitive to immunotherapy. However, immunotherapy is currently only approved for endometrial cancer if the cancer has come back after receiving chemotherapy.

Tislelizumab is an experimental drug. This means that it has not been approved for use by the regulatory agencies (FDA) in the US, but it has been approved in China. Tislelizumab is a monoclonal antibody acting on a protein called Programmed Cell Death 1 (PD-1). In this study, we would like to study how a new immunotherapy (tislelizumab (BGB-A317) works for patients who have not yet received chemotherapy and how the tumor and the immune system respond to treatment.


### 2. How many people will take part in this study?

10-20 patients in total will be enrolled at The Ohio State University.

### 3. What will happen if I take part in this study?

### Before you begin the study:

You will need to sign this informed consent form.

You will need to have the following exams, tests or procedures to find out if you can be in the study. These exams, tests or procedures are part of regular cancer care and may be done even if you do not join the study. If you have had some of them recently, they may not need to be repeated. This will be up to your study doctor.

- 1. History and physical examination will include blood pressure measurement and weight and pelvic examination to evaluate if there is tumor growing in your pelvis or vagina.
- 2. Blood tests to assess blood cell counts; liver, kidney and blood clotting function; blood mineral levels; CA-125 levels (marker in your blood to monitor your cancer if this has been a marker for you).
- 3. Hepatitis testing for hepatitis B virus and hepatitis C virus. If a test shows you have an active hepatitis B or C infection, you will have follow-up counselling and medical advice provided by the Institution. If your test results are positive, the study doctors may be required by law to notify government health authorities. Signing the consent form means that you agree to have this testing; it will not be done without your consent.
- 4. Urine test sample for urine protein level and a pregnancy test if you could become pregnant.
- 5. If you are able to become pregnant, a blood test will be done to make sure that you are not pregnant.
- 6. Electrocardiogram (EKG)
- 7. Computed tomography [CT] scan will be obtained prior to treatment of your chest, abdomen and pelvis to determine where your tumor is located, and to determine the size of the tumor.
- 8. An eye exam by an appropriate specialist. This will include a visual acuity test, which is used to determine the smallest letters you can read on a standardized eye chart, and optical coherence tomography, or equivalent, which is a noninvasive technique used for examining the retina. These exams are useful in diagnosing eye conditions. If eye exams cannot be performed at the same location as the study site and the patient requires eye exam(s) be performed at other eye clinics or other hospitals, your doctor may recommend you have the eye exam(s) performed at


another eye clinic or other hospital. Please discuss the details regarding these arrangements with your doctor.

- 9. Patients who are suspected or known to have serious respiratory concurrent illness or exhibit significant respiratory symptoms unrelated to underlying cancer should take a pulmonary function test
- 10. If your doctor has additional concerns that the study medication may not be safe for you, you may require additional tests to confirm you are a good candidate for the study (for example, if you have a history of significant and/or uncontrolled heart problems you may need an ultrasound of your heart).

If the exams, tests and procedures show that you can be in the study, and you choose to take part, you will proceed with the study.

### Biopsy

Your tumor will be tested using a sample of your tumor tissue from either a previous or recent surgery or biopsy. If you do not have tissue available, you will need to have a biopsy in order to obtain a sample of tissue. A biopsy may require taking a small sample of your tumor tissue; either with the use of a large needle (incisional or core biopsy) or with surgical forceps (forceps biopsy). Alternatively, a small sample of your tumor may be removed by cutting it out surgically (excisional biopsy), or with a special round-shaped knife (punch biopsy). The biopsy procedure you may have depends on the location and accessibility of your tumor. Your study doctor will explain the details of this procedure to you.

#### **During the study:**

- 1. History and physical examination every 3 weeks on day 1 of every cycle which will include blood pressure measurement and may include pelvic examination.
- 2. Eye exam will be repeated every 15 weeks (approximately every 5 cycles)
- 3. CT scan or MRI scan after the first 9 weeks and if your tumor is improving then you will have imaging studies approximately every 9 weeks (3 cycles). If your doctor suspects that your cancer is growing you will also get imaging studies.
- 4. Periodic blood testing for CA-125 level if you have ovarian cancer or if you have endometrial cancer and your CA-125 is initially elevated. CA-125 is a blood test that is generally performed for patients with your type of cancer to monitor the effectiveness of treatment.
- 5. Blood tests to assess blood cell counts; liver and kidney function; blood mineral levels prior to day 1 of every cycle to make sure your body has recovered and it is safe to get chemotherapy. Your bloodwork will include thyroid function test every other cycle
- 6. Toxicity Assessments that involve asking you details about side effects of treatment will occur on day 1, 8, 15of cycle 1 and day 1 of each cycle after that.
- 7. You are not allowed to take steroids while on this study. Please check with your doctor before taking steroids.


#### Treatment:

You will receive immunotherapy with tislelizumab (BGB A317).

<u>Tislelizumab</u> is given through a vein (intravenously/IV) every 3 weeks. Throughout the study you will be monitored closely for side effects. The initial infusion (Cycle 1 Day 1) will be delivered over 60 minutes. If tislelizumab is well tolerated, then the subsequent infusions may be administered over 30 minutes, which is shortest amount of time that is allowed for administering the infusion. As a routine precaution after each infusion, you will be monitored for a period of 30 minutes.

You will have routine chemotherapy visits every 3 weeks (on day 1 of each 3-week cycle) with your gynecologic oncologist and intravenous immunotherapy on the same day for as long as you are on this treatment.

Your chemotherapy is given as an outpatient and your outpatient visit (including seeing your doctor) will take 2-3 hours. You can continue to be on this treatment as long as you are receiving benefit (cancer is shrinking or cancer is not growing and you are feeling well).

After cycle 1 (day 7-21 after your first treatment) you will have a biopsy to see how the immunotherapy is affecting the tumor.

After the first three cycles you will also get imaging to see how well the treatment is working.

If your cancer has not gone away after 3 cycle of immunotherapy and you have not previously received chemotherapy, we will add 2 standard chemotherapy agents (carboplatin and paclitaxel) to see if we can improve the treatment response (make the cancer shrink more or resolve).

You will have another biopsy after you receive the 3 drug combination to study if and how the immunotherapy with chemotherapy is affecting your tumor.

Whether you are on just immunotherapy or the combination of standard chemotherapy and immunotherapy, we will do imaging every 3 cycles (9 weeks) for the first year of therapy. After the first year, we will do imaging every 12 weeks. You will always have the option to go off trial if you do not demonstrate a complete response and can start cytotoxic chemotherapy (carboplatin/paclitaxel or other chemotherapy) or enroll on another clinical trial.

After 6-9 cycles of tislelizumab/carboplatin/paclitaxel, you may continue single agent tislelizumab maintenance every 3 weeks for a total of 24 months as long as you are


receiving benefit (cancer is shrinking or cancer is not growing and you are feeling well).

If you have previously received chemotherapy, tislelizumab may be continued for 24 months, as long as you are receiving benefit (cancer is shrinking or cancer is not growing and you are feeling well).

If the cancer continues to grow and does not improve with treatment you will have a biopsy to study why the immunotherapy (with or without chemotherapy) is not working for your tumor.

If you decide to stop taking this treatment, or your doctor decides to stop treatment because your cancer starts growing back, you will be monitored for side effects for 30 days after stopping treatment those 30 days. You will have your normal cancer follow up visits. You will not need to fill out any additional surveys or paperwork since all information will be collected from the medical records. If you continue follow up or treatment with a different doctor or hospital, we may contact you periodically (every 3-6 months) to see how you are doing.



Studies that are not part of standard of care:


**Blood samples:** You will be asked to give extra blood samples before your first treatment and before cycle 2, 3, 4, 6, 9, 12, and at the time of cancer progression or stopping treatment. This blood test would not be needed for diagnosis but helps to study how your body and the treatment work to fight your cancer. No more than 10 teaspoons (about 46mL) of blood will be collected at one time.

**Tissue Specimens:** To better understand which patients are more likely to benefit from this treatment, we will be asking you to allow us to collect and store some tissue for research. You will need 3-4 research biopsies during this study. The tissue collected will not be needed for diagnostic purposes but will be used to study how the immunotherapy affects your tumor and why it works or why it does not work. If you have any other biopsies during or after the study, or have already existing specimens (from a previous surgery or biopsy) that are no longer needed for your care, we may study these as well.

**Clinical Data:** We are asking you to allow us to collect and store clinical data from your medical record for research. This includes data about your surgery and specimens collected, treatment plans, pathology and cytology reports, and genetic testing, if performed.


| | Screening | Treatment Cycles | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Assessment | | Cycles 1 to 3<br>(Every 21 days) | | | Cycle 4 and<br>Subsequent<br>Cycles<br>(Every 21 Days) | End-of-Treatment<br>Visit | Safety Follow-up | Survival<br>Follow-up |
| Days (Window) | -28 to ~ -1 | 1 (± 3) | 8 (± 2) | 15 (± 2) | 1 (± 3) | 0 to 7 Days | 30 ± 7 Days After<br>Last Dose | Every 3<br>Months |
| Informed consent | Х | | | | | | | |
| Demographics/medical<br>history/prior medications | х | | | | | | | |
| Vital signs, Physical Exam,<br>performance status, height,<br>weight, | х | х | | | х | Х | х | |
| Eye Exams | Х | | | | Х | χ | Х | |
| Toxicity Assessments | Х | Х | Х | Х | Х | Х | Х | Х |
| Concomitant medications | Х | Х | Х | Х | Х | Х | Х | |
| Safety Blood & Urine Labs | Х | х | Х | Х | Х | χ | Х | |
| Pregnancy test | Х | | | | Х | Х | Х | |
| Pulmonary function tests | Х | | | | Х | χ | Х | |
| Research Blood | Х | | | | Х | Х | | |
| Imaging | х | Every 9 weeks for the first 52 weeks, then every 12 weeks after 52 weeks until disease progression or removal from study | | | | | | |
| Tumor Tissue/Biopsy | Х | Х | | Х | Х | Х | | |
| Tislelizumab administration | | х | | | Х | | | |
| Carboplatin/paclitaxel | | | | | Х | | | |
| Electrocardiogram (12-Lead) | Х | | | | | Х | | |
| Survival visits/phone calls | | | | | | | | |

## During the study you will not be allowed to take

- Other chemotherapy or supplements that could treat cancer
- Live vaccines within 30 days prior to the first dose of study treatment and while
  participating in the study. Examples of live vaccines include, but are not
  limited to, the following: measles, mumps, rubella, varicella/zoster, yellow
  fever, rabies, BCG, and typhoid vaccine. Seasonal influenza vaccines for
  injection are generally killed virus vaccines and are allowed; however,


intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.

- Steroids unless your doctor approves this.
- Any other medications that can interfere or interact with the study treatments.
  These can make the cancer treatment work too much or too little resulting in
  side effects. Always check with your doctor if new medications are allowed
  (even if prescribed for a short duration)

### 4. How long will I be in the study?

You may stop your participation in the study at any time.

You can stay on the study as long as you are doing well and your cancer has not gotten worse. If you are doing well on treatment and your cancer is not getting worse, treatment will continue if you and your study doctor agree to this. If you are not tolerating treatment well and/or your cancer is getting worse, treatment will stop. After you finish treatment, you will need to return to the clinic 30 days following the last dose of treatment to make sure you have recovered from any side effects. You will also be asked what anti-cancer therapy you may be getting. If you cancer grows while on study you will be offered to biopsy the tumor again. This biopsy is for research only in order to study why your cancer may have become

If your cancer has not gotten worse or has resolved, then you will need to return to the clinic at the time your treating physician recommends (usually every 8-12 weeks). Imaging will be done if your doctor believes this is indicated. You may be contacted by the study staff every 3-4 months to see how you are and to find out what anticancer therapy you may be getting for the year after completing study treatment.

#### 5. Can I stop being in the study?

resistant to the treatment.

You may leave the study at any time. If you decide to stop participating in the study, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. Your decision will not affect your future relationship with The Ohio State University.

# 6. What risks, side effects or discomforts can I expect from being in the study?

<u>Physical Risks:</u> When you have a test or procedure to remove tissue for your standard of care, your doctor will explain the risks at that time, and they may include discomfort, bleeding, bruising, and scarring. You may experience discomfort, bleeding or bruising associated with the blood draw and/or biopsy.


<u>Privacy Risks:</u> Every effort will be made to maintain your privacy, however this cannot be guaranteed. There is a risk in this project that someone other than researchers could get access to information we have stored about you. If that data suggested something serious about your health, it could be misused.

Research using your specimens may include mapping your DNA (whole genome sequencing). This information could identify you. Ask the study team if you have questions.

#### **GINA**

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions about your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information from this research when making a decision to hire, promote, or fire you or when setting the terms of your employment.

All health insurance companies and group health plans must follow this federal law. This law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Under Ohio law, health insurance companies cannot ask about the results of a genetic test or use any information obtained from genetic testing to make decisions about providing coverage or benefits for health care services.

### General / Unforeseeable

You may have side effects while on the study. Everyone taking part in the study will be watched carefully for any side effects. However, doctors don't know all the side effects that may happen. Side effects may be mild or very serious. Your health care team may give you medicines to help lessen side effects. Many side effects go away soon after you stop taking lenvatinib, pembrolizumab and paclitaxel. In some cases, side effects can be serious in that they can be long lasting, may never go away, may result in hospitalization, or may be life threatening and possibly lead to death (fatal).

You should talk to your study doctor about any side effects that you have while taking part in the study.

#### **Risks Associated With Tislelizumab**

Tislelizumab is an investigational agent that is currently in clinical development. It is FDA approved in China, but not in the US at this time. Limited safety data are


available in patients and the full safety profile has not been characterized. The following recommendation is based on results from nonclinical and clinical studies with tislelizumab and published data on other molecules within the same biologic class.

The PD-L1/PD-1 pathway is involved in peripheral immune tolerance; therefore, such therapy may increase the risk of immune related side effects, specifically the induction or enhancement of autoimmune conditions.

The study treatment may affect how different parts of your body work, such as your liver, kidneys, heart, and blood. The study doctor will be testing your blood and will let you know if changes occurred that may affect your health. Tislelizumab, and other drugs similar to tislelizumab, are thought to act against cancer by activating the immune system to attack cancer. However, in some patients, there can be side effects related to an over-active immune system, which can cause damage to your organs or other tissues of your body. In most cases, these side effects are temporary and can be treated with stopping tislelizumab and treating you with a medication that suppresses the immune system (for example, steroids).

### Side effects known to be associated with tislelizumab as a single agent

The effects of tislelizumab on humans are not yet fully known. Tislelizumab is an investigational drug that has only been administered to a limited number of patients in clinical studies. As of 20 May 2020, 1,328 patients have received at least 1 dose of tislelizumab as a single agent.

The most commonly reported side effects seen in patients taking tislelizumab as a single agent are outlined below. In most cases, these side effects are mild and respond to treatment, but in some cases may be serious or require urgent treatment. Some of these side effects may be life-threatening or fatal.

# Very common side effects (occurring in at least 1 out of 10 people; equal to or more than 10.0%).

- Nausea (feeling sick to the stomach)
- Constipation
- Diarrhea (watery, loose, or soft stools)
- Fever
- Fatigue (tiredness)
- Vomiting
- Abnormal liver function measured by liver tests (blood aspartate aminotransferase increased, alanine aminotransferase increased, or bilirubin increased, which may reflect liver damage)Rash
- Itching
- Anemia


- Decreased appetite
- Cough
- Underactive thyroid gland (possible feeling cold, weight gain, heart failure, and/or constipation)

# Common (occurring in at least 1 out of 100 and less than 1 out of 10; equal to or more than 1.0% but less than 10.0%).

- Inflammation of the mouth and lips
- Inflammation of the large bowel
- Chills
- Blood alkaline phosphatase increased (abnormal liver test; possible liver damage)
- High blood sugar (possible diabetes)
- Thrombocytopenia (abnormally low levels of a blood cells called platelets or thrombocytes; this can interfere with your ability to stop bleeding when you are injured)
- Low level of white blood cells in the blood (can interfere with your ability to fight infection)
- Low level of neutrophils in the blood (a type of white blood cell that fights infection)
- High blood sugar
- Shortness of breath, Lung inflammation (possible difficulty breathing)
- Overactive thyroid gland (possible weight loss, heart rate changes, and/or sweating)
- Inflammation of the thyroid gland (possible tenderness in the neck)
- Joint pain
- Muscle pain
- Headache
- Dizziness
- Inflammation of the liver (also called hepatitis)


Abnormal liver function

Reaction to the injection of tislelizumab (also called an infusion-related reaction; may happen soon after the injection; symptoms include flushing, difficulty breathing, feeling faint, chills, itching, and/or skin rash)

Uncommon serious side effects (occurring in at least 1 out of 1,000 and less than 1 out of 100 people; equal to or more than 0.1% but less than 1.0%).

- Inflammation of the pancreas
- Severe skin reaction
- Abnormally low level of lymphocytes in the blood (lymphocytes are a white blood cell with important functions in the immune system)
- Diabetes mellitus
- Decreased production of adrenal hormones (also known as stress hormones; can lead to weakness and/or low blood pressure)
- Arthritis (joint inflammation and swelling)
- Muscle inflammation
- Inflammation of the heart muscle (usually caused by infection; may be serious and require hospitalization)
- Inflammation inside the eye

#### Kidney inflammation

# Risks Associated with Tislelizumab in Combination with Chemotherapy (carboplatin and paclitaxel)

As of 20 May 2020, a total of 54 patients have taken part in this open label combination study. In addition to the side effects listed above for tislelizumab as a single agent, the following side effects for this combination observed in ≥ 5% of patients and assessed as related to tislelizumab by an Investigator are listed below.

# Very common side effects (occurring in at least 1 out of 10 people; equal to or more than 10.0%).

- Asthenia (weakness)
- Hypothyroidism (underactive thyroid gland [possible weight gain, heart failure, and/or constipation])


# Common side effects (occurring in at least 1 out of 100 and less than 1 out of 10 people; equal to or more than 1.0% but less than 10.0%).

- Blood thyroid stimulating hormone increased (underactive thyroid gland [possible weight gain, heart failure, and/or constipation])
- Alpha hydroxybutyrate dehydrogenase increased (abnormal blood test)
- Blood creatine phosphokinase increased (increased blood level of enzyme from muscle)
- Proteinuria (excess protein in the urine. This may cause fluid retention)

# <u>Possible Side Effects of Carboplatin</u> (CTEP Table Version Date: October 23, 2018)

## **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Carboplatin, more than 20 and up to 100 may have:

- Infection, especially when white blood cell count is low
- Bruising, bleeding
- Anemia which may cause tiredness, or may require blood transfusions
- Vomiting, nausea
- Pain
- Hair loss

## OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Carboplatin, from 4 to 20 may have:

- Visual loss
- Diarrhea, Constipation, belly pain
- Changes in taste
- Numbness and tingling in fingers and toes

#### RARE, AND SERIOUS

In 100 people receiving Carboplatin, 3 or fewer may have:

 Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat

# <u>Possible Side Effects of Paclitaxel</u> (CTEP Table Version Date: September 26, 2017)

### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving Paclitaxel, more than 20 and up to 100 may have:

- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Infection, especially when white blood cell count is low
- Bruising, bleeding
- Anemia which may cause tiredness, or may require blood transfusions


#### COMMON, SOME MAY BE SERIOUS

In 100 people receiving Paclitaxel, more than 20 and up to 100 may have:

- Pain
- Sores in mouth which may cause difficulty swallowing
- Diarrhea, nausea, vomiting
- Muscle weakness
- Numbness, tingling or pain of the arms and legs
- Hair loss

#### OCCASIONAL. SOME MAY BE SERIOUS

In 100 people receiving Paclitaxel, from 4 to 20 may have:

- Abnormal heartbeat
- Blood clot which may cause swelling, pain, shortness of breath
- Damage to the lungs which may cause shortness of breath

#### RARE, AND SERIOUS

In 100 people receiving Paclitaxel, 3 or fewer may have:

- Heart attack or heart failure which may cause shortness of breath, swelling of ankles, and tiredness
- A tear or a hole in the bowels which may cause pain or that may require surgery
- Severe skin rash with blisters and peeling which can involve mouth and other parts of the body

**Other medications:** There are certain medications and supplements that may interact with the study drug(s). You should not take any new medications or supplements without discussing it with your study doctor first.

**Blood samples:** Collection of treatment related and research related blood samples: Taking blood from your arm may sometimes cause pain/discomfort at the site where the blood is drawn, bruising, bleeding, occasional lightheadedness, redness, and/or swelling, and, rarely, faintness or infection.

**Biopsies:** Collection of research biopsies may cause pain or discomfort at the site and can cause damage to the tissue and surrounding tissues or organs.

For more information about risks and side effects, ask your study doctor.

Precautions will be taken to try to prevent side effects from occurring, and medicines are available to treat many side effects if they do occur. For example, you may


develop signs of an allergic reaction during any given treatment with paclitaxel, pembrolizumab or lenvatinib, which could be severe or life threatening. The symptoms of the allergic reaction may include rash, sweating, swelling of the skin, itching, change in heart rate, difficulty breathing, low blood pressure and abdominal, back, arm or leg pain.

If these symptoms develop, you will be treated promptly with medications to control the allergic reaction. You may need to be put into the hospital if the allergic reaction becomes severe or life threatening. Before any treatment with paclitaxel, you will receive medications prior to each treatment to try to prevent an allergic reaction.

## Reproductive Risks

You should not become pregnant while on this study because the drug(s) in this study can affect an unborn baby. Women should not breastfeed while on this study. It is important you understand that if you could become pregnant, you need to use birth control while on this study. Check with your study doctor about what kind of birth control methods to use and how long to use them. Some methods might not be approved for use in this study. You should notify your health care team immediately if you think you have become pregnant while participating in this study.

## **Imaging Risks**

The CT scans that you get in this study to monitor if your cancer has responded to treatment will expose you to low amounts of radiation. Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. This type of radiation is called "background radiation." No one knows for sure whether exposure to these low amounts of radiation is harmful to your body.

As part of the CT scans that you get in this study, you will get oral contrast to drink and iodine will be injected into your vein. Some people are allergic to iodine. Let your study doctor know if you have an allergy to iodine or seafood or if you have kidney problems.

### 6. What benefits can I expect from being in the study?

You may potentially benefit from your cancer shrinking or disappearing because of the chemotherapy. However, no direct medical benefit can be guaranteed. No promise can be made concerning the study outcome because results from a clinical research study cannot be predicted. The benefit of the study to society may be the use of information gained why this treatment works or does not work on certain tumors so we can better predict which patients may benefit from this treatment in the future.


## 7. What other choices do I have if I do not take part in the study?

You may choose not to participate without penalty or loss of benefits to which you are otherwise entitled. Your decision to not participate in the study will not affect your treatment. Should you decide to decline this study, your gynecologic oncologist will discuss the possibility of other treatments such as other chemotherapy or best supportive care.

## 8. What are the costs of taking part in this study?

The Study Drug, Tislelizumab will be provided by the sponsor. You and your insurance company will not be billed for this study drug while you are on the study. Also, all procedures that are required only for this study, and that are not part of your regular medical care, will not be billed to you or your insurance.

You or your insurance company will need to pay for medicines and clinic, hospital, and doctors' services that are part of your regular medical care.

Participating in this research study may lead to additional costs to you. In some cases, it is possible that your insurance company will not pay for these costs because you are taking part in a research study. You will be responsible for any co-payments, co-insurance, and/or deductibles as required by your insurance company.

For more information on clinical trials and insurance coverage, you can visit the National Cancer Institute's Web site at <a href="http://cancer.gov/clinicaltrials/understanding/insurance-coverage">http://cancer.gov/clinicaltrials/understanding/insurance-coverage</a>. You can print a copy of the "Clinical Trials and Insurance Coverage" information from this Web site.

Another way to get the information is to call 1-800-4-CANCER (1-800-422-6237) and ask them to send you a free copy.

## 9. Will I be paid for taking part in this study?

You will not receive any compensation for participating in this study. The institution receives payment from Beigene that covers some but not all of the costs of the study. This payment helps pay for paperwork involved in study. It does not pay you or your caregivers for taking part in this study.

If you agree to participate, your samples will be considered a gift to The Ohio State University. The university may sell or share your samples and personal information with others, such as private companies, government agencies, or other universities. The university will be paid if your samples and personal information are sold.


 Your samples and personal information may be used to make new products or technologies. You will not be paid if these new products or technologies are sold or make money.

 You cannot choose how your samples and personal information will be used. If you do not want to let others decide how your samples and personal information will be used, then you should not donate your samples.

#### 10. What happens if I am injured because I took part in this study?

If you suffer an injury from participating in this study, you should notify the researcher or study doctor immediately, who will determine if you should obtain medical treatment at The Ohio State University Wexner Medical Center.

The cost for this treatment will be billed to you or your medical or hospital insurance. The Ohio State University has no funds set aside for the payment of health care expenses for this study.

### 11. What are my rights if I take part in this study?

If you choose to participate in the study, you may discontinue participation at any time without penalty or loss of benefits. By signing this form, you do not give up any personal legal rights you may have as a participant in this study.

You will be provided with any new information that develops during the course of the research that may affect your decision whether or not to continue participation in the study.

You may refuse to participate in this study without penalty or loss of benefits to which you are otherwise entitled.

An Institutional Review Board responsible for human subjects research at The Ohio State University reviewed this research project and found it to be acceptable, according to applicable state and federal regulations and University policies designed to protect the rights and welfare of research participants.

## 12. Will my de-identified information (and bio-specimens) be used or shared for future research

Yes, it/they may be used or shared with other researchers without your additional informed consent.


## 13. Will my study-related information be kept confidential?

Efforts will be made to keep your study-related information confidential. However, there may be circumstances where this information must be released. For example, personal information regarding your participation in this study may be disclosed if required by state law.

Also, your records may be reviewed by the following groups (as applicable to the research):

- Office for Human Research Protections or other federal, state, or international regulatory agencies;
- U.S. Food and Drug Administration;
- The Ohio State University Institutional Review Board or Office of Responsible Research Practices;
- The sponsor supporting the study, their agents or study monitors; and
- Your insurance company (if charges are billed to insurance).
- Natera/Signatera

Data stored will consist data that has been collected as part of your normal care and is part of your medical records. Any additional testing will be for research only and will not be shared with you.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search the website at any time.

## 14. HIPAA AUTHORIZATION TO USE AND DISCLOSE INFORMATION FOR RESEARCH PURPOSES

#### I. What information may be used and given to others?

- · Past and present medical records;
- Research records;
- Records about phone calls made as part of this research;
- Records about your study visits;
- Information that includes personal identifiers, such as your name, or a number associated with you as an individual;
- Information gathered for this research about:


HIV / AIDS

Hepatitis infection

Sexually transmitted diseases

Other reportable infectious diseases

Physical exams

Laboratory, x-ray, and other test results

Diaries and questionnaires

The diagnosis and treatment of a mental health condition

- Records about any study drug you received;
- · Records about the study device; and

### II. Who may use and give out information about you?

Researchers and study staff.

#### III. Who might get this information?

- The sponsor of this research. "Sponsor" means any persons or companies that are:
  - working for or with the sponsor (for example Natera/Signatera for research samples); or
  - owned by the sponsor.
- Authorized Ohio State University staff not involved in the study may be aware that you are participating in a research study and have access to your information;
- If this study is related to your medical care, your study-related information may be placed in your permanent hospital, clinic, or physician's office record;
- Others: data safety monitoring boards

#### IV. Your information may be given to:

- The U.S. Food and Drug Administration (FDA), Department of Health and Human Services (DHHS) agencies, and other federal and state entities;
- Governmental agencies in other countries;
- Governmental agencies to whom certain diseases (reportable diseases) must be reported; and
- The Ohio State University units involved in managing and approving the research study including the Office of Research and the Office of Responsible Research Practices.

### V. Why will this information be used and/or given to others?


- To do the research;
- To study the results; and
- To make sure that the research was done right.

#### VI. When will my permission end?

There is no date at which your permission ends. Your information will be used indefinitely. This is because the information used and created during the study may be analyzed for many years, and it is not possible to know when this will be complete.

#### VII. May I withdraw or revoke (cancel) my permission?

Yes. Your authorization will be good for the time period indicated above unless you change your mind and revoke it in writing. You may withdraw or take away your permission to use and disclose your health information at any time. You do this by sending written notice to the researchers. If you withdraw your permission, you will not be able to stay in this study. When you withdraw your permission, no new health information identifying you will be gathered after that date. Information that has already been gathered may still be used and given to others.

## VIII. What if I decide not to give permission to use and give out my health information?

Then you will not be able to be in this research study and receive research-related treatment. However, if you are being treated as a patient here, you will still be able to receive care.

#### IX. Is my health information protected after it has been given to others?

There is a risk that your information will be given to others without your permission. Any information that is shared may no longer be protected by federal privacy rules.

#### X. May I review or copy my information?

Signing this authorization also means that you may not be able to see or copy your study-related information until the study is completed.

#### 15. Who can answer my questions about the study?


For questions, concerns, or complaints about the study, or if you feel you have been harmed as a result of study participation, you may contact Dr. Floor Backes or Kelly Dodd at 614-366-9084.

For questions related to your privacy rights under HIPAA or related to this research authorization, please contact Privacy Officer, Suite E2140, 600 Ackerman Road, Columbus, OH 43202, 614-293-4477.

For questions about your rights as a participant in this study or to discuss other study-related concerns or complaints with someone who is not part of the research team, you may contact the Office of Responsible Research Practices at 1-800-678-6251.

If you are injured as a result of participating in this study or for questions about a study-related injury, you may contact Dr. Floor Backes or Kelly Dodd RN at (614) 366-9084


## Signing the consent form

I have read (or someone has read to me) this form and I am aware that I am being asked to participate in a research study. I have had the opportunity to ask questions and have had them answered to my satisfaction. I voluntarily agree to participate in this study.

I am not giving up any legal rights by signing this form. I will be given a copy of this combined consent and HIPAA research authorization form.

| | Printed name of participant | Signature of participant | |
|---|---|---|---|
| | | A | M/PM |
| | | Date and time | |
| | Printed name of person authorized to consent for participant (when applicable) | Signature of person authorized to consent for participant (when applicable) | to |
| | Relationship to the participant | Date and time | M/PM |
| <u>าv</u> | estigator/Research Staff | | |
| ha<br>eq | estigator/Research Staff ave explained the research to the particip uesting the signature(s) above. There are form has been given to the participant o | e no blanks in this document. A copy | / of |
| ha<br>eq | ave explained the research to the particip uesting the signature(s) above. There ar | e no blanks in this document. A copy | / of |
| ha<br>eq | eve explained the research to the particip uesting the signature(s) above. There are form has been given to the participant o | e no blanks in this document. A copy r his/her representative. Signature of person obtaining consent | / of |


| Witness(es) - May be left blank if no | ot required by the IRB | |
|---------------------------------------|------------------------|-------|
| Printed name of witness | Signature of witness | |
| | Date and time | AM/PM |
| Printed name of witness | Signature of witness | |
| | Date and time | AM/PM |